CLINICAL TRIAL: NCT07194174
Title: Effect of Physical Training in Individuals With Hypokalemic and Hyperkalemic Periodic Paralysis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Annica Buss Enegaard, BSc, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-25003151
Record Dates: First submitted 2025-09-10; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Hypokalemic Periodic Paralysis; Hyperkalemic Periodic Paralysis
MeSH Terms: conditions — Hypokalemic Periodic Paralysis; Paralysis, Hyperkalemic Periodic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hypo-/HyperPP (Experimental): Strength exercise will be implemented for all participants included in this study. The first 12 weeks will be without intervention and after this period the intervention will begin. The participants are therefore all controls (no intervention) and experimental (intervention).
  Interventions: Other: Strength exercise

INTERVENTIONS:
Other: Strength exercise — 3 weekly supervised trainings with specific strengt exercises

SUMMARY:
This study wishes to investigate the effects of strength exercise in patients with either HypoPP or HyperPP.

The investigators wishes to include participants already diagnosed with either HypoPP or HyperPP in af 24 week prospective study where the patients will be tested and asked to fill out questionnaires three times. These appointments will be schedueled at week 0, week 12 and week 24.

In the time period between week 12 and week 24, the patients will have a personalized strength exercise program, which they will have to follow these 3 months. The exercise will be supervised by one or more of the investigators.

ELIGIBILITY:
Inclusion Criteria:

* Patients with genetic verified HypoPP or HyperPP
* Age minimum 18 years
* Able to walk a minimum of 10 meters independently with or without assistive devices and be able to stand from a chair without using hands

Exclusion Criteria:

* Other significant cause of muscle weakness
* Heart or lung disease which, in the investigator's opinion, makes participation in the study training inadvisable

Exclusion from muscle biopsy

* Anticoagulant treatment
* Impaired blood clotting due to disease

Exclusion from MRI scanning due to:

* Metal implants in the body that contraindicate MRI scanning or are positioned such that the scan quality is significantly affected
* Claustrophobia
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Functional endurance test in the form of the Five Times Sit-to-Stand Test (5STS) | From intervention to end of intervention at 12 weeks

SECONDARY OUTCOMES:
Functional endurance test in the form of the 6-Minute Walk Test (6MWT) | 12 weeks
Muscle strength measured with a dynamometer | 12 weeks
  Dynamometer used: Biodex
Number of attacks of muscle weakness | 12 weeks
  Self-reported by participants
Myotonia graded using the Myotonia Behaviour Scale (MBS) | 12 weeks
  Scale goes from 0-5, where 0 is no stiffness and 5 is incapacitating stiffness, which demands constant movement to not be totally locked up
Quality of life measured with the Individualized Neuromuscular Quality of Life Questionnaire (INQoL) | 12 weeks
  To assess health-related quality of life of patient suffering from neuromuscular diseases.
Quality of life measured with the EuroQol 5 Dimensions 5 Levels (EQ-5D-5L) | 12 weeks
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflects the patient's own judgement.
Fatigue measured with the Multidimensional Fatigue Inventory (MFI-20) | 12 weeks
  A questionnaire consisting of 20 questions. The higher the collected score upon answering all the questions indicates a more severe fatigue.
Pain graded using the Visual Analog Scale (VAS) | 12 weeks
  A pain scale from 0-10, where 0 is no pain and 10 is the worst pain possible

IPD SHARING:
Plan to Share IPD: No